CLINICAL TRIAL: NCT06089486
Title: Multiparametric Cardiac Positron Emission Tomography for Cardiac Allograft Vasculopathy Surveillance After Heart Transplantation
Brief Title: MARINER Trial: Multiparametric Cardiac PET for CAV Surveillance After Heart Transplantation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Heart Institute Research Corporation (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 20230460-01T
Record Dates: First submitted 2023-09-29; First posted 2023-10-18 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Cardiac Allograft Vasculopathy
Keywords: Heart Transplant

STUDY DESIGN:
Intervention Model Description: 1:1 randomization to PET or ICA
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Invasive Coronary Angiography (Other): Patients in this arm will undergo annual CAV surveillance with ICA
  Interventions: Diagnostic Test: ICA
- Positron Emission Tomography (Other): Patients in this arm will undergo annual CAV surveillance with PET
  Interventions: Diagnostic Test: PET

INTERVENTIONS:
Diagnostic Test: ICA — Patients will undergo annual CAV surveillance with ICA
  Arms: Invasive Coronary Angiography
Diagnostic Test: PET — Patients will undergo annual CAV surveillance with PET
  Arms: Positron Emission Tomography

SUMMARY:
Cardiac allograft vasculopathy (CAV) is a common complication affecting heart transplant patients. This condition causes narrowing of the heart arteries leading to graft dysfunction. Surveillance for CAV is vital; however an ideal approach has not been established. The goal of this study is to assess whether noninvasive positron emission tomography (PET) based surveillance is non-inferior to invasive coronary angiography (ICA) surveillance.

DETAILED DESCRIPTION:
MARINER is a Canadian multicentre prospective, randomized clinical outcomes-based trial evaluating noninferiority of a noninvasive PET strategy compared to ICA for CAV surveillance. Patients are randomized to annual PET or ICA for CAV surveillance. Non-inferiority is assessed according to a clinical composite of death, retransplant, allograft dysfunction not related to acute rejection, and angiographic CAV associated with myocardial infarction or heart failure. Secondary outcomes include the rate of new or progressive CAV, number of ICA performed, number of ICA and PET procedural related complications, EuroQol-5 Dimension assessed patient health-related quality of life and health care resource use.

ELIGIBILITY:
Inclusion Criteria:

1. Post heart transplant 2-10 years.
2. Age ≥18 years.
3. Able to provide informed consent.

Exclusion Criteria:

1. Contraindication to dipyridamole due to severe aortic stenosis.
2. Contraindication to dipyridamole due to 2:1 or greater AV block without pacemaker.
3. Contraindication to dipyridamole due to severe bronchospasm.
4. Unable to undergo coronary angiography due to allergy to iodinated contrast.
5. Unable to undergo coronary angiography due to glomerular filtration rate ≤30 mL/min/1.73 m2. for non-dialysis patients as determined by local laboratory analysis.
6. Unable to undergo coronary angiography due to unsuitable vascular access.
7. Treated rejection ≤1-month.
8. Unstable angina or MI ≤7 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 576 (Estimated)
Dates: Start 2024-01-08 (Actual); Primary Completion 2028-10 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
Clinically relevant composite: Death | From date of randomization up to a minimum of 2 years
  Date of death due to any cause
Clinically relevant composite: Retransplant | From date of randomization up to a minimum of 2 years
  Heart retransplantation for any indication
Clinically relevant composite: Allograft Dysfunction | From date of randomization up to a minimum of 2 years
  ≥25% decrease in left ventricular ejection fraction
Clinically relevant composite: CAV with Heart Failure or Myocardial Infarction | From date of randomization up to a minimum of 2 years
  Angiographic evidence of CAV (ISHLT CAV 1-3)

SECONDARY OUTCOMES:
Rate of new or progressive CAV | From date of randomization up to a minimum of 2 years
  CAV disease severity according to ISHLT CAV 0-3 grading and/or MIT on IVUS
Number of ICA performed | From date of randomization up to a minimum of 2 years
  Number of ICA performed for any indication including CAV surveillance, abnormal PET or clinical indication
Number of procedural related complications (ICA and PET) | From date of randomization up to a minimum of 2 years
  The frequency of ICA and PET procedural related complication including vascular access complications, stroke, MI, arrhythmia, drug allergy and contrast nephropathy
Patient Health related outcomes | Baseline and 12-monthly up to a minimum of 2 years
  EuroQol-5 Dimension is a standardized health related questionnaire measuring 5 domains of health and a state of health using a visual analog scale (best state marked 100 and worst state marked 0)
Health Resource Utilization | From date of randomization up to a minimum of 2 years
  Cost effectiveness of each CAV surveillance strategy (ICA and PET)

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Chih, Principal Investigator — Ottawa Heart Institute Research Corporation
Locations (5):
- Canada (5):
  - University of Calgary, Calgary, Alberta
  - Mazankowski Alberta Heart Institute, Edmonton, Alberta
  - University of Ottawa Heart Institute, Ottawa, Ontario
  - Toronto-General Hospital - University Health Network, Toronto, Ontario
  - Montreal Heart Institute, Montreal, Quebec